CLINICAL TRIAL: NCT06827418
Title: The Effect of Simulation and Peer Teaching Methods on Nursing Students' Assessment of Blood Pressure: A Randomised Controlled Trial
Brief Title: The Effect of Simulation and Peer Teaching Methods on Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Evrim Eyikara, Gazi University Faculty of Nursing, doctoral assistant professor, Gazi University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: E.1156965
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure; Simulation Training; Peer Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer teaching (Experimental): Experimental Group 1 (Peer Teaching): Students will practice the psychomotor steps of blood pressure measurement through peer teaching. Third- and fourth-year nursing students will serve as peer educators. Students will apply the skill steps under the guidance of an upper-class peer instructor.
- simulation (Experimental): Experimental Group 2 (Simulation): Students will practice the psychomotor steps of blood pressure measurement using a simulator.
  Interventions: Other: simulation
- control group (No Intervention): Control Group (Traditional Laboratory Training): Students will practice the psychomotor steps of blood pressure measurement through traditional laboratory training, which is instructor-centered. They will practice blood pressure measurement steps on low-fidelity mannequins and on each other.

INTERVENTIONS:
Other: simulation — Students will practice the psychomotor steps of blood pressure measurement using a simulator.
  Arms: simulation
Other: peer teaching — Students will practice the psychomotor steps of blood pressure measurement through peer teaching. Third- and fourth-year nursing students will serve as peer educators. Students will apply the skill steps under the guidance of an upper-class peer instructor.

SUMMARY:
The aim of this study is to determine the effect of simulation and peer teaching methods on nursing students' ability to assess blood pressure. The study population will consist of first-year nursing students. All students will complete the "Demographic Characteristics Form" and the "Blood Pressure Knowledge Test" (pre-test). Students will be randomized according to their average scores, and three groups will be formed. Experimental Group 1 Students will practice the psychomotor steps of blood pressure measurement through peer teaching. Experimental Group 2 students will practice the psychomotor steps of blood pressure measurement using a simulator. Control group students will practice the psychomotor steps of blood pressure measurement through traditional laboratory training, which is instructor-centered. They will practice blood pressure measurement steps on low-fidelity mannequins and on each other. After completing the two-session psychomotor skills training, all students will be assessed using the "VAS" to determine their confidence and anxiety levels. One week after the training, all students will measure the blood pressure of a healthy adult in the skills laboratory. During the measurement, the researcher will evaluate the students using the "Blood Pressure Measurement Checklist." After the procedure, the students will complete the "Blood Pressure Knowledge Test" (post-test) and the "VAS" to assess their confidence and anxiety levels. Four to six weeks after the training, all students will measure the blood pressure of a hospitalized adult patient in a clinical setting. Following the procedure, students will complete the "Blood Pressure Knowledge Test" (floow up test) and the "VAS" (third measurement) to assess their confidence and anxiety levels.

DETAILED DESCRIPTION:
Deficiencies in basic skills pose a significant threat to patient safety. Therefore, the training, practice, and evaluation components of basic skills such as blood pressure measurement should be renewed as needed. Simulation is a teaching method that allows students to practice in a realistic and safe environment, enabling repetition without the risk of causing harm. Simulation is particularly important in nursing education due to the increasing number of students, the insufficient number of educators, its accessibility and repeatability in learning opportunities, and its role in ensuring patient safety. Another effective method frequently used in teaching blood pressure measurement in nursing education is peer teaching. It defines a collaborative teaching and learning strategy. Peer teaching is a relational process in which a more experienced individual contributes to the professional and personal development of a less experienced individual. In peer teaching, students can ask their peers questions without hesitation, benefit from a stress-free learning environment, and experience increased academic success through mutual support. As a result, it can improve nursing students' academic performance and enhance the retention rates of nursing courses.

The aim of this study is to determine the effect of simulation and peer teaching methods on nursing students' ability to assess blood pressure. The study population will consist of first-year nursing students who will enroll in the Fundamentals of Nursing course at Gazi University Faculty of Nursing during the spring semester of the 2024-2025 academic year. Based on a power analysis conducted using the GPower 3.1.9.7 program, the sample size was determined to be 28 participants per group, with a total of 84 participants, considering a Type 1 error of 0.05, a Type 2 error of 0.20, and an effect size of f = 0.35 for detecting differences in measurements between groups. Considering possible dropouts, the sample size was increased by 10%, and a total of 93 participants (31 per group) will be included in the study.

Data collection tools will include the "Demographic Characteristics Form," "Blood Pressure Knowledge Test," "Blood Pressure Measurement Checklist," and "Visual Analog Scale (VAS)." During the spring semester of the 2024-2025 academic year, theoretical lectures on blood pressure measurement will be conducted within the Fundamentals of Nursing course. Researchers will demonstrate blood pressure measurement techniques and show a video illustrating the skill steps. All students will complete the "Demographic Characteristics Form" and the "Blood Pressure Knowledge Test" (pre-test). Then, students who voluntarily agree to participate will be selected based on inclusion criteria. Students will be randomized according to their average scores, and three groups will be formed. Each group will be taught blood pressure psychomotor skills using different instructional methods. The training for each group will be conducted in different laboratories simultaneously.

* Experimental Group 1 (Peer Teaching): Students will practice the psychomotor steps of blood pressure measurement through peer teaching. Third- and fourth-year nursing students will serve as peer educators. Students will apply the skill steps under the guidance of an upper-class peer instructor.
* Experimental Group 2 (Simulation): Students will practice the psychomotor steps of blood pressure measurement using a simulator.
* Control Group (Traditional Laboratory Training): Students will practice the psychomotor steps of blood pressure measurement through traditional laboratory training, which is instructor-centered. They will practice blood pressure measurement steps on low-fidelity mannequins and on each other.

After completing the two-session psychomotor skills training, all students will be assessed using the "VAS" (first measurement) to determine their confidence and anxiety levels.

One week after the training, all students will measure the blood pressure of a healthy adult in the skills laboratory. Each student will perform the procedure individually. During the measurement, the researcher will evaluate the students using the "Blood Pressure Measurement Checklist." The observing instructor will mark each checklist item as "observed," "incorrect/incomplete," or "not observed." After the procedure, the students will complete the "Blood Pressure Knowledge Test" (post-test) and the "VAS" (second measurement) to assess their confidence and anxiety levels.

Four to six weeks after the training, all students will measure the blood pressure of a hospitalized adult patient in a clinical setting. Each student will perform the procedure individually. The researcher will evaluate the students using the "Blood Pressure Measurement Checklist," while the observing instructor will mark each item on the checklist as "observed," "incorrect/incomplete," or "not observed." Following the procedure, students will complete the "Blood Pressure Knowledge Test" (retention test) and the "VAS" (third measurement) to assess their confidence and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* First-time enrollment in the Fundamentals of Nursing course
* Willingness to participate in the study

Exclusion Criteria:

* Having a high school, associate degree, or bachelor's degree in a health-related field
* Having previously taken a course on blood pressure measurement
* Having a hearing impairment
* The student choosing to withdraw from the study at any stage
* Failure to complete the data collection forms

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Cognitive knowledge related to blood pressure | from enrollment to the end of the 6-week follow-up period.
  The Blood Pressure Knowledge Test will be used for assessment. It was developed by Takmak and Kurban (2018) and consists of 20 multiple-choice questions, each with five options. Each question has only one correct answer.
blood pressure psychomotor measurement skill | from the teaching methods are applied to the end of the 6-week follow-up period
  The Blood Pressure Measurement Checklist will be used for assessment. It consists of procedural steps that thoroughly evaluate the process of blood pressure measurement and assessment. To ensure an objective evaluation of students, it has been designed as a rubric-based scoring tool. The checklist is categorized as follows: **"Correct" (2 points), "Incorrect/Incomplete" (1 point), and "Not Observed" (0 points).**
confidence and anxiety levels | from the teaching methods are applied to the end of the 6-week follow-up period
  The Visual Analog Scale (VAS) will be used for assessment. It is a single-item measurement tool that allows participants to mark their subjective state on a visual scale, providing a simple and quick application. The scale is typically a 100 mm horizontal line, on which participants indicate their perceived level. As the score increases, confidence level and anxiety level also increase.**

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Sarıtaş, Principal Investigator — doctor research assistant
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No